CLINICAL TRIAL: NCT00119600
Title: A Randomised, Multi-Center, Double-Blind, Placebo-Controlled, Dose-Finding Study of AMG 114 Administered by Subcutaneous Injection for the Treatment of Anemia in Subjects With Non-Myeloid Malignancies Receiving Multicycle Chemotherapy
Brief Title: A Study of AMG 114 Administered by Subcutaneous Injection for the Treatment of Anemia in Subjects With Non-Myeloid Malignancies Receiving Multicycle Chemotherapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20030205
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2009-05-11 (Estimated); Status verified 2009-05

CONDITIONS: Anemia; Cancer
Keywords: Non-myeloid malignancy; Clinical Trial
MeSH Terms: conditions — Anemia; Neoplasms

INTERVENTIONS:
Drug: AMG 114

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of AMG 114 administered subcutaneously for the treatment of chemotherapy induced anemia in subjects receiving multicycle chemotherapy.

ELIGIBILITY:
Inclusion Criteria: Part A: - Non-myeloid malignancy receiving multicycle chemotherapy - Receiving non-platinum containing chemotherapy - At least 6 additional weeks of cyclic cytotoxic chemotherapy planned Part B and Part C: - Non-myeloid malignancy receiving multicycle chemotherapy - At least 12 additional weeks of cyclic cytotoxic chemotherapy planned All Parts: - Chemotherapy induced anemia - Greater than 6 month life expectancy - ECOG 0-2 - Adequate renal and liver function Exclusion Criteria: - Chronic myeloid leukemia, AML, ALL, Burkitt's lymphoma or lymphoblastic lymphoma - History of seizure disorder - Primary hematologic disorder which could cause anemia, other than a non-myeloid malignancy - Unstable angina, congestive heart failure or uncontrolled cardiac arrhythmia - Uncontrolled hypertension - History of pure red cell aplasia - Clinically significant inflammatory disease or active infection - Iron deficiency - ANC less than 0.8 x 10^9 cells/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Incidence and severity of adverse events
Change in hemoglobin concentration
Maximum observed concentration (Cmax)
Time Cmax is observed (Tmax)
AUC

SECONDARY OUTCOMES:
Change in FACT-fatigue sub-scores

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_59_AMG_114_20030205.pdf